CLINICAL TRIAL: NCT03706209
Title: A Phase II, Multicenter, Double-blind, Placebo-controlled, Efficacy and Safety Trial of Two Oral Doses (150 mg Bid / 300 mg Bid) of MP1032 in Male and Female Patients With Moderate-to-Severe Chronic Plaque Psoriasis
Brief Title: Study to Evaluate Efficacy and Safety of MP1032 in Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MetrioPharm AG (Industry)
Collaborators: Bioskin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP1032-CT04; 2017-003484-36 (EudraCT Number)
Record Dates: First submitted 2018-10-04; First posted 2018-10-15 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis
Keywords: moderate to severe; chronic; plaque psoriasis
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome | interventions — sodium luminolate

STUDY DESIGN:
Intervention Model Description: Three-arm randomized, double-blind, placebo-controlled, parallel group phase II multi-center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 150 mg MP1032 bid (Experimental): 3 × 50 mg (150 mg) MP1032 plus 3 × placebo hard gelatin capsules (per dosage) are provided twice daily over a period of 12 weeks.
  Interventions: Drug: MP1032; Drug: Placebo
- 300 mg MP1032 bid (Experimental): 6 × 50 mg (300 mg) MP1032 hard gelatin capsules (per dosage) are provided twice daily over a period of 12 weeks.
  Interventions: Drug: MP1032
- Placebo bid (Placebo Comparator): 6 × placebo hard gelatin capsules (per dosage) are provided twice daily over a period of 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP1032 — hard gelatin capsules containing 50mg MP1032 as active ingredient
  Arms: 150 mg MP1032 bid; 300 mg MP1032 bid
Drug: Placebo — hard gelatin capsules containing no active ingredient
  Arms: 150 mg MP1032 bid; Placebo bid

SUMMARY:
The primary objective of this trial is to evaluate the clinical efficacy and safety of two oral doses of MP1032 (150 mg bid and 300 mg bid) when taken for 12 weeks by patients with moderate-to-severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, parallel, placebo-controlled trial to evaluate the efficacy and safety of two oral doses of MP1032 (150 mg bid and 300 mg bid) in adult patients with moderate-to-severe chronic plaque psoriasis.

The trial design consists of a 28-day screening period, a 12-week treatment period, and subsequently a 28-day follow-up period. Each patient will have 6 visits and unscheduled visits as needed.

Approximately 150 patients (2 × 50 patients MP1032 and 50 patients placebo) who meet the entry criteria will be randomized on Day 1 to receive either 150 mg MP1032, 300 mg MP1032 or placebo orally twice daily for 12 weeks. The administration of IMP will stop after end of study (in max. 13 weeks).

PASI (Psoriasis Area and Severity Index), PGA (Physician Global Assessment) and BSA (Body Surface Area) Scores will be recorded at predefined timepoints as basis for the efficacy evaluation.

Safety parameter will be monitored from the signing of the informed consent form (ICF) until the last follow-up visit.

To evaluate systemic concentrations of MP1032 PK (pharmacokinetics) samples will be analyzed in a subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent.
2. Adult male and female patients between 18 years and 70 years with moderate-to-severe chronic plaque psoriasis (diagnosed by Investigator):

   1. PASI score ≥10 - ≤20 at baseline
   2. BSA score: > 10%
   3. Stable disease duration of ≥ 6 months at the initiation of IMP.
   4. topical therapy fails to control the disease
3. Body Mass Index (BMI) between 18.5 and 34.9 kg/m2.
4. Women of childbearing potential (WCBP) must have a negative serum pregnancy test at Screening (Visit 1). In addition, sexually active WCBP must agree to use adequate contraception throughout the trial (see Section 3.2 for more details on adequate contraception):

   1. A method with less than 1% failure rate OR
   2. Abstinence
5. Post-menopausal women with spontaneous amenorrhea for at least 12 months and women on hormonal replacement therapy (HRT). The use of hormonal replacement therapy (HRT) during the trial is permitted, however for these patients an appropriate contraception method according to Inclusion Criterion 4 must be ensured. Sterilized women may be included (see Section 3.2 for more details on sterile definition)
6. Male patients who are sexually active with a female partner and are not surgically sterile (vasectomy performed at least six months prior to treatment) must agree to inform their female sexual partner to use an acceptable form of birth control as described in the informed consent form. For females, an acceptable method (Pearl Index < 1%) would be to use implants, injectable, combined oral contraceptives, some intrauterine devices, or be postmenopausal, be surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy)
7. In good health as judged by the investigator, based on medical history, physical examination, serum chemistry, hematology and urinalysis
8. Patients must meet the following clinical laboratory criteria:

   * White blood cell count ≥3.5 × 109/L
   * Platelet count ≥100 × 109/L
   * Serum creatinine ≤1.5 × upper limit of normal (ULN); estimated glomerular filtration rate >60 mL/min
   * Total bilirubin ≤1.5 × ULN
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN
   * Hemoglobin ≥ lower limit of normal as per central laboratory reference ranges for women and men accordingly
   * No coagulopathy (International Normalized Ratio [INR] <1.5)
9. Patients agree to minimize normal sun exposure during the course of the trial
10. Patients are considered reliable and capable of adhering to the protocol (e.g. able to understand the patient information and complete diaries), visit schedule, or medication intake according to the judgment of the Investigator.

Exclusion Criteria:

1. Patients with non-plaque form of psoriasis (erythrodermic, guttate, pustular form of psoriasis). Associated psoriasis arthritis is allowed provided no other in-/exclusion criteria are influenced, no forbidden concomitant therapy is required for the well -being of the patient and there is no impact on trial objectives as determined by the Investigator.
2. Treatment with concomitant medication that may affect and provoke or aggravate psoriasis, e.g. antimalarial drugs, beta-blockers or ACE (angiotensin-converting-enzyme) inhibitors unless on a stable dose for 3 months before IMP intake.
3. Evidence of skin conditions at the time of Screening Visit other than psoriasis that would interfere with evaluations of the effect of the IMP on psoriasis.
4. Patients with any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the ICF, as assessed by the investigator.
5. Pregnant or lactating women or women planning to become pregnant during the trial and / or within 28 days following the last dose of IMP.
6. Male patients planning a partner pregnancy or sperm donation during the trial including follow up period.
7. Known allergies to any ingredient of the IMP e.g. mannitol, macrophage modulators, or gelatin.
8. History or symptoms of a clinically significant illness in the four weeks before first treatment and during the trial that in the opinion of the investigator may place the patient at risk by trial participation or influence the outcome of the trial. Well controlled diseases such as hypertension, hyperlipidemia, diabetes or hypothyroidism are permitted.
9. Patients with active malignancy or history of malignancy, except for basal cell and actinic keratosis. Basal cell carcinoma of the skin or in situ cervical carcinoma that have been fully treated and show no evidence of recurrence are allowed.
10. Positive HIV-Antibody, HBs-Antigen or HCV-Antibody-Test at screening.
11. Previous strong sun exposure (e.g. sea holiday) within 28 days or UV treatment within 24 weeks before IMP initiation.
12. Known photo allergy and / or experienced drug-induced photo toxicity.
13. Elective (planned) hospitalization or medical intervention preventing patient from following the protocol requirements.
14. Prior treatment not adhering to defined drug classes and related washout periods (Protocol table 2.)
15. Planned use of any ultraviolet (UV) phototherapy or photochemotherapy / photosensitizing drugs during the course of the trial and within 28 days/24 weeks following the last dose of the IMP.
16. Patients with a history of chronic alcohol or drug abuse within 6 months of IMP initiation.
17. Patients with a blood pressure outside the given range of 160 mm Hg (systolic) and 95 mm Hg (diastolic)
18. Patients who are employed by MetrioPharm, contract research organization (CRO) or clinical site involved in the clinical trial.
19. Vulnerable patients (e.g. patients kept in detention).
20. Patients who are unable to communicate, read or understand the local language, or who display another condition, which, in the Investigator's opinion, makes them unsuitable for clinical trial participation.
21. Patient is institutionalized because of legal or regulatory order.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (10):
  - Dr. Tsianakas / Dr. Ameluxen, Bad Bentheim
  - Rothaar Studien GmbH, Berlin
  - Dr. Johannes Niesmann / Dr. Othlinghaus, Bochum
  - Klinische Forschung Dresden GmbH, Dresden
  - MensingDerma, Hamburg
  - MVZ DermaKiel, Kiel
  - Hautarztpraxis Dres. med. Scholz, Sebastian, Schilling, Mahlow
  - Universitätsmedizin Mainz, Hautklinik und Poliklinik, Mainz
  - Klinische Forschung Schwerin (kfsn), Schwerin
  - Centroderm GmbH, Wuppertal
- Poland (9):
  - GynCentrum Sp. Z o.o., Katowice
  - MULTIKLINIKA SALUTE Sp. z o. o., Katowice
  - Provita Sp. z o.o., Centrum Medyczne Angelius Provita, Katowice
  - CENTRUM MEDYCZNE PLEJADY Sp. z o. o. spółka komandytowa, Krakow
  - Dermoklinika Centrum Medyczne s.c. M.Kierstan, J.Narbutt, A.Lesiak, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Kliniczny Szpital Wojewódzki nr 1 im. Fryderyka Chopina w Rzeszowie, Klinika Dermatologii, Rzeszów
  - Laser Clinic s.c. Andrzej Królicki, Tomasz Kochanowski, Szczecin
  - DermMEDICA Sp. z o.o., Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 150 mg MP1032 Bid: 3 × 50 mg (150 mg) MP1032 plus 3 × placebo hard gelatin capsules (per dosage) provided twice daily over a period of 12 weeks.
  MP1032: hard gelatin capsules containing 50mg MP1032 as active ingredient
  Placebo: hard gelatin capsules containing no active ingredient
- 300 mg MP1032 Bid: 6 × 50 mg (300 mg) MP1032 hard gelatin capsules (per dosage) provided twice daily over a period of 12 weeks.
  MP1032: hard gelatin capsules containing 50mg MP1032 as active ingredient
- Placebo Bid: 6 × placebo hard gelatin capsules (per dosage) provided twice daily over a period of 12 weeks.
  Placebo: hard gelatin capsules containing no active ingredient
Period: Overall Study
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Started | 52 | 48 | 55
Completed | 36 | 39 | 39
Not Completed | 16 | 9 | 16

BASELINE CHARACTERISTICS:
Population: The safety-evaluation-set (SES) included all patients that were randomized and received any trial medication at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid | Total
Number analyzed (Participants) | 51 | 48 | 55 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 48 | 46 | 52 | 146
  >=65 years | 3 | 2 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 20 | 48
  Male | 41 | 30 | 35 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 51 | 48 | 55 | 154
  other | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 39 | 34 | 40 | 113
  Germany | 12 | 14 | 15 | 41

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 - Week 12 (EoT)
Description: Percentage of patients reaching PASI 75 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 75% in the PASI score at End-of-Treatment (EoT) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: The full-analysis-set (FAS) included all randomized patients who received at least one dose of IMP and had at least one post-baseline assessment. The FAS was considered primary analysis set for the efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 4 | 4 | 1
  Non-Responder | 46 | 43 | 53
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.161, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.12, 95% CI 2-sided [0.47 to 35.97]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.111, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.52, 95% CI 2-sided [0.55 to 55.43]

2. Primary Outcome: PGA Improvement - Week 12 (EoT)
Description: PGA improvement rate in treatment groups (150 and 300 mg bid) compared to placebo. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The number of responders corresponds to the number of patients with an improvement of 1 or more points on the 7-points PGA scale at End-of-Treatment (EoT) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 14 | 14 | 10
  Non-Responder | 36 | 33 | 44
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.222, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.71 to 4.25]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.182, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.75 to 4.91]

3. Secondary Outcome: PASI 75 VCS - Week 12 (EoT)
Description: Percentage of patients reaching PASI 75 in treatment groups (150 and 300 mg bid) compared to placebo in the valid cases set (VCS). The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 75% in the PASI score at End-of-Treatment (EoT) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: The valid-cases-set (VCS) included all patients from the full-analysis-set (FAS), who completed the assessment of the co-primary endpoints without any protocol violation interfering with the precise evaluation of treatment efficacy and with sufficient exposure to IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 32 | 36 | 34
Participants
  Responder | 3 | 3 | 1
  Non-Responder | 29 | 33 | 33
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.294, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.91, 95% CI 2-sided [0.33 to 25.39]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.291, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.06, 95% CI 2-sided [0.31 to 53.14]

4. Secondary Outcome: PGA Improvement VCS - Week 12 (EoT)
Description: PGA improvement rate in treatment groups (150 and 300 mg bid) compared to placebo in the valid-cases-set (VCS). The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The number of responders corresponds to the number of patients with an improvement of 1 or more points on the 7-points PGA scale at End-of-Treatment (EoT) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 32 | 36 | 34
Participants
  Responder | 9 | 13 | 8
  Non-Responder | 23 | 23 | 26
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.617, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.45 to 3.77]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.319, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.6 to 5]

5. Secondary Outcome: PASI 50 - Week 12 (EoT)
Description: Percentage of patients reaching PASI 50 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 50% in the PASI score at End-of-Treatment (EoT) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 8 | 10 | 6
  Non-Responder | 42 | 37 | 48
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.47, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.5 to 4.52]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.136, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.44, 95% CI 2-sided [0.76 to 7.82]

6. Secondary Outcome: PASI ANCOVA Change From Baseline - Week 12 (EoT)
Description: Mean PASI score and change to baseline in treatment groups (150 and 300mg) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. Displayed are changes in the PASI score (LS mean estimates) at end of treatment (EoT) compared to baseline in the different arms in patients of the FAS subject analysis set wherein negative values indicate a better outcome.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale (PASI baseline change)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI baseline change) | 0.1 (1.0) | -1.1 (1.0) | -0.1 (1.0)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.894, ANCOVA; least square means = 0.2, 95% CI 2-sided [-2.6 to 3], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Estimates and treatment comparison of least square means using an ANCOVA model, with treatment arm and (pooled) analysis center as factors and baseline outcome as covariate; Test type: Superiority; p = 0.456, ANCOVA; least square means = -1.1, 95% CI 2-sided [-3.8 to 1.7], Standard Error of Mean 1.4

7. Secondary Outcome: PASI Descriptive Statistics - Week 12 (EoT)
Description: Mean PASI score and change to baseline in treatment groups (150 and 300mg) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. For the change of baseline negative values indicate improvement and positive values indicate worsening.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (PASI)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI)
  Day 1 | 14.7 (2.8) | 14.2 (2.7) | 13.8 (2.5)
  Week 12 (EoT) | 15 (9.1) | 13 (9) | 13.5 (6)
  Week 12 (EoT) - change from baseline | 0.3 (8.4) | -1.2 (7.6) | -0.3 (5.5)

8. Secondary Outcome: Time to PASI 75
Description: Time to the achievement of PASI 75, if applicable. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. Displayed is the number of responders that reached an improvement of at least 75% in the PASI score in the respective week.
Time Frame: from treatment start (Study Day 1 - Baseline) to either Study Day 25, 56, 84 (EoT) or 112 (FU)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Week 4 | 0 | 1 | 2
  Week 8 | 2 | 0 | 0
  Week 12 (EoT) | 3 | 3 | 1
  Week 16 (FU) | 0 | 2 | 1
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.572, Log Rank; Kaplan-Meier estimate of the median time (day) to reach the PASI 75 criterion was not computed since data were too sparse
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.4494, Log Rank; [statistical method as in outcome 8, analysis 1]

9. Secondary Outcome: Time to PASI 50
Description: Time to the achievement of PASI 50, if applicable. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies. It is a physician's assessment of psoriasis that is a therapeutic standard in clinical studies for this disease. Displayed is the number of responders that reached an improvement of at least 50% in the PASI score in the respective week.
Time Frame: from treatment start (Study Day 1 - Baseline) to either Study Day 25, 56, 84 (EoT) or 112 (FU)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Week 4 | 2 | 7 | 5
  Week 8 | 4 | 3 | 2
  Week 12 (EoT) | 4 | 3 | 2
  Week 16 (FU) | 1 | 3 | 2
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.7922, Log Rank; Kaplan-Meier estimate of the median time (day) to reach the PASI 50 criterion was not computed since data were too sparse
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.1425, Log Rank; [statistical method as in outcome 9, analysis 1]

10. Secondary Outcome: PGA Descriptive Statistics - Week 12 (EoT)
Description: Mean PGA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at end of treatment. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). For change from baseline negative values indicate improvement.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (PGA)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PGA)
  Day 1 | 4.1 (0.7) | 4.2 (0.7) | 4.1 (0.7)
  Week 12 (EoT) | 4.0 (1.3) | 3.8 (1.2) | 4.1 (1.0)
  Week 12 (EoT) - change from baseline | -0.1 (1.1) | -0.4 (1.0) | -0.0 (0.8)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.992, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.143, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0

11. Secondary Outcome: PGA Frequency Counts - Week 12 (EoT)
Description: The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The 7-point's assessment of psoriasis is a therapeutic standard in clinical studies for this disease. Frequency of the scores from 0 to 6 at end of treatment in the different treatment groups is displayed.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 1 | 1 | 0
  2 - Mild | 6 | 7 | 4
  3 - Mild to Moderate | 10 | 9 | 11
  4 - Moderate | 15 | 15 | 18
  5 - Moderate to Severe | 12 | 13 | 18
  6 - Severe | 6 | 2 | 3

12. Secondary Outcome: BSA Descriptive Statistics - Week 12 (EoT)
Description: Mean BSA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at end of treatment. The BSA (Body Surface Area) provides information on the total surface area of the body affected with psoriasis plaques in percent (%).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
percentage of body surface area
  Day 1 | 19 (8.8) | 19.2 (10.5) | 17.5 (6.3)
  Week 12 (EoT) | 20.2 (13) | 19.7 (17.2) | 17.3 (8.7)
  Week 12 (EoT) - change from baseline | 1.2 (9.4) | 0.5 (11.3) | -0.2 (5.3)

13. Secondary Outcome: PASI 75 - Week 4
Description: Percentage of patients reaching PASI 75 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 75% in the PASI score at the respective visit (week 4) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 0 | 1 | 2
  Non-Responder | 50 | 46 | 52
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.178, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.718, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.63, 95% CI 2-sided [0.05 to 7.48]

14. Secondary Outcome: PASI 75 - Week 8
Description: Percentage of patients reaching PASI 75 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 75% in the PASI score at the respective visit (week 8) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 2 | 1 | 1
  Non-Responder | 48 | 46 | 53
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.474, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.4, 95% CI 2-sided [0.21 to 28.05]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.867, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.08 to 19.05]

15. Secondary Outcome: PASI 75 - Week 16 (FU)
Description: Percentage of patients reaching PASI 75 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 75% in the PASI score at the respective visit (Follow Up) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
Participants
  Responder | 4 | 5 | 2
  Non-Responder | 34 | 35 | 42
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.375, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.38 to 12.84]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.116, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.24, 95% CI 2-sided [0.66 to 27.08]

16. Secondary Outcome: PASI 50 - Week 4
Description: Percentage of patients reaching PASI 50 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 50% in the PASI score at the respective visit (week 4) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 2 | 7 | 5
  Non-Responder | 48 | 40 | 49
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.287, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.41, 95% CI 2-sided [0.08 to 2.27]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.332, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.53 to 6.4]

17. Secondary Outcome: PASI 50 - Week 8
Description: Percentage of patients reaching PASI 50 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 50% in the PASI score at the respective visit (week 8) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 5 | 9 | 7
  Non-Responder | 45 | 38 | 47
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.719, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.25 to 2.63]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.357, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.72, 95% CI 2-sided [0.55 to 5.32]

18. Secondary Outcome: PASI 50 - Week 16 (FU)
Description: Percentage of patients reaching PASI 50 in treatment groups (150 and 300 mg bid) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. The number of responders corresponds to the number of patients with an improvement of at least 50% in the PASI score at the respective visit (Follow Up) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
Participants
  Responder | 8 | 10 | 6
  Non-Responder | 30 | 30 | 38
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.355, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.53 to 5.72]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.198, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.22, 95% CI 2-sided [0.67 to 7.37]

19. Secondary Outcome: PASI ANCOVA Change From Baseline - Week 4
Description: Mean PASI score and change to baseline in treatment groups (150 and 300mg) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. Displayed are changes in the PASI score (LS mean estimates) at the respective visit (week 4) compared to baseline in the different arms in patients of the FAS subject analysis set wherein negative values indicate a better outcome.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale (PASI baseline change)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI baseline change) | -0.3 (0.7) | -1.7 (0.7) | -0.6 (0.7)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.757, ANCOVA; least square means = 0.3, 95% CI 2-sided [-1.7 to 2.3], Standard Error of Mean 1
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.267, ANCOVA; least square means = -1.1, 95% CI 2-sided [-3.1 to 0.9], Standard Error of Mean 1

20. Secondary Outcome: PASI ANCOVA Change From Baseline - Week 8
Description: Mean PASI score and change to baseline in treatment groups (150 and 300mg) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies with a maximum value of 72 points, any value higher than 10 is considered as moderate to severe psoriasis. It is a physician's assessment of psoriasis that is a therapeutic standard in clinical studies for this disease. Displayed are changes in the PASI score (LS mean estimates) at the respective visit (week 8) compared to baseline in the different arms in patients of the FAS subject analysis set wherein negative values indicate a better outcome.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale (PASI baseline change)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI baseline change) | 0.2 (0.9) | -1.8 (0.9) | -0.8 (0.8)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.412, ANCOVA; least square means = 1, 95% CI 2-sided [-1.4 to 3.4], Standard Error of Mean 1.2
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.401, ANCOVA; least square means = -1, 95% CI 2-sided [-3.5 to 1.4], Standard Error of Mean 1.2

21. Secondary Outcome: PASI ANCOVA Change From Baseline - Week 16 (FU)
Description: Mean PASI score and change to baseline in treatment groups (150 and 300mg) compared to placebo. The PASI (psoriasis area severity index) is the most commonly used and validated assessment for grading the severity of psoriasis in clinical studies and combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease) wherein any value higher than 10 is considered as moderate to severe psoriasis. Displayed are changes in the PASI score (LS mean estimates) at the respective visit (week 16, FU) compared to baseline in the different arms in patients of the FAS subject analysis set wherein negative values indicate a better outcome.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale (PASI baseline change)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
score on a scale (PASI baseline change) | -0.3 (1.3) | -0.8 (1.2) | -0.8 (1.2)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.801, ANCOVA; least square means = 0.4, 95% CI 2-sided [-3 to 3.9], Standard Error of Mean 1.7
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; [analysis description as in outcome 6, analysis 2]; Test type: Superiority; p = 0.957, ANCOVA; least square means = 0.1, 95% CI 2-sided [-3.4 to 3.3], Standard Error of Mean 1.7

22. Secondary Outcome: PASI Descriptive Statistics - Week 4
Description: as for outcome 7
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (PASI)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI)
  Day 1 | 14.7 (2.8) | 14.2 (2.7) | 13.8 (2.5)
  Week 4 | 14.5 (7.1) | 12.4 (5.5) | 13.1 (4.6)
  Week 4 - change from baseline | -0.2 (6.3) | -1.8 (4.2) | -0.7 (4.1)

23. Secondary Outcome: PASI Descriptive Statistics - Week 8
Description: as for outcome 7
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (PASI)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
score on a scale (PASI)
  Day 1 | 14.7 (2.8) | 14.2 (2.7) | 13.8 (2.5)
  Week 8 | 15.1 (8.1) | 12.3 (7.8) | 12.8 (5.4)
  Week 8 - change from baseline | 0.4 (7.4) | -1.9 (6.4) | -1 (4.9)

24. Secondary Outcome: PASI Descriptive Statistics - Week 16 (FU)
Description: as for outcome 7
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale (PASI)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
score on a scale (PASI)
  Week 16 (FU) | 15.1 (9.3) | 13.6 (11) | 12.3 (5.1)
  Week 16 (FU) - change from baseline | 0.3 (9) | -0.7 (9.6) | -1.2 (4.7)

25. Secondary Outcome: PGA Improvement - Week 4
Description: PGA improvement rate in treatment groups (150 and 300 mg bid) compared to placebo. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The number of responders corresponds to the number of patients with an improvement of 1 or more points on the 7-points PGA scale at the respective visit (week 4) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 11 | 13 | 9
  Non-Responder | 39 | 34 | 45
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.45, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.55 to 3.8]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.186, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.97, 95% CI 2-sided [0.74 to 5.26]

26. Secondary Outcome: PGA Improvement - Week 8
Description: PGA improvement rate in treatment groups (150 and 300 mg bid) compared to placebo. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The number of responders corresponds to the number of patients with an improvement of 1 or more points on the 7-points PGA scale at the respective visit (week 8) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  Responder | 12 | 16 | 14
  Non-Responder | 38 | 31 | 40
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.884, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.41 to 2.18]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.384, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.61 to 3.64]

27. Secondary Outcome: PGA Improvement - Week 16 (FU)
Description: PGA improvement rate in treatment groups (150 and 300 mg bid) compared to placebo. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). The number of responders corresponds to the number of patients with an improvement of 1 or more points on the 7-points PGA scale at the respective visit (Follow Up) compared to baseline.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
Participants
  Responder | 14 | 13 | 12
  Non-Responder | 24 | 27 | 32
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.311, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.63 to 4.26]
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.699, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.47 to 3.17]

28. Secondary Outcome: PGA Descriptive Statistics - Week 4
Description: Mean PGA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at the respective visit (week 4). The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PGA score
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
PGA score
  Day 1 | 4.1 (0.7) | 4.2 (0.7) | 4.1 (0.7)
  Week 4 | 3.9 (0.9) | 3.9 (0.9) | 4.0 (1.0)
  Week 4 - change from baseline | -0.1 (0.7) | -0.3 (0.6) | -0.1 (0.6)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.671, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.183, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0

29. Secondary Outcome: PGA Descriptive Statistics - Week 8
Description: Mean PGA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at the respective visit (week 8). The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PGA score
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
PGA score
  Day 1 | 4.1 (0.7) | 4.2 (0.7) | 4.1 (0.7)
  Week 8 | 4.0 (1.1) | 3.8 (1.1) | 3.9 (1.1)
  Week 8 - change from baseline | -0.1 (0.9) | -0.4 (0.8) | -0.2 (0.8)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.542, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.328, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0

30. Secondary Outcome: PGA Descriptive Statistics - Week 16 (FU)
Description: Mean PGA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at Follow Up visit. The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: PGA score
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
PGA score
  Day 1 | 4.1 (0.7) | 4.2 (0.7) | 4.1 (0.7)
  Week 16 (FU) | 3.8 (1.3) | 3.8 (1.3) | 3.9 (1.1)
  Week 16 (FU) - change from baseline | -0.2 (1.1) | -0.4 (1.1) | -0.1 (0.7)
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.921, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.488, Wilcoxon (Mann-Whitney); Hodges-Lehmann using location shift = 0, 95% CI 2-sided [0 to 0], Standard Error of Mean 0

31. Secondary Outcome: PGA Frequency Counts - Day 1 (Baseline)
Description: The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). Frequency of different scores at the respective visit (baseline) is displayed.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 0 | 0 | 0
  2 - Mild | 1 | 0 | 0
  3 - Mild to Moderate | 8 | 8 | 11
  4 - Moderate | 28 | 24 | 27
  5 - Moderate to Severe | 13 | 14 | 15
  6 - Severe | 0 | 1 | 1

32. Secondary Outcome: PGA Frequency Counts - Week 4
Description: The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). Frequency of different scores at the respective visit (week 4) is displayed.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 0 | 0 | 0
  2 - Mild | 2 | 2 | 5
  3 - Mild to Moderate | 15 | 13 | 10
  4 - Moderate | 19 | 21 | 20
  5 - Moderate to Severe | 12 | 10 | 19
  6 - Severe | 2 | 1 | 0

33. Secondary Outcome: PGA Frequency Counts - Week 8
Description: The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). Frequency of different scores at the respective visit (week 8) is displayed.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
Participants
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 0 | 1 | 1
  2 - Mild | 5 | 5 | 6
  3 - Mild to Moderate | 11 | 11 | 10
  4 - Moderate | 17 | 18 | 17
  5 - Moderate to Severe | 14 | 9 | 19
  6 - Severe | 3 | 3 | 1

34. Secondary Outcome: PGA Frequency Counts - Week 16 (FU)
Description: The PGA (Physician's global assessment) provides an overall evaluation of the severity of the disease ranging from 0 (clear skin - no diseases) to 6 (severe disease). Frequency of different scores at follow up visit is displayed.
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
Participants
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 2 | 3 | 1
  2 - Mild | 4 | 4 | 4
  3 - Mild to Moderate | 10 | 8 | 10
  4 - Moderate | 9 | 11 | 14
  5 - Moderate to Severe | 10 | 12 | 13
  6 - Severe | 3 | 2 | 2

35. Secondary Outcome: BSA Descriptive Statistics - Week 4
Description: Mean BSA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at the respective visit (week 4). The BSA (Body Surface Area) provides information on the total surface area of the body affected with psoriasis plaques in percent (%).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
percentage of body surface area
  Day 1 | 19 (8.8) | 19.2 (10.5) | 17.5 (6.3)
  Week 4 | 19.7 (12.4) | 18.3 (11.9) | 17.1 (7.1)
  Week 4 - change from baseline | 0.7 (8.3) | -0.9 (6.3) | -0.4 (3.1)

36. Secondary Outcome: BSA Descriptive Statistics - Week 8
Description: Mean BSA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at the respective visit (week 8). The BSA (Body Surface Area) provides information on the total surface area of the body affected with psoriasis plaques in percent (%).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 50 | 47 | 54
percentage of body surface area
  Day 1 | 19 (8.8) | 19.2 (10.5) | 17.5 (6.3)
  Week 8 | 20.4 (12.9) | 18.6 (14.7) | 16.6 (7.9)
  Week 8 - change from baseline | 1.4 (9.5) | -0.6 (9) | -0.9 (3.9)

37. Secondary Outcome: BSA Descriptive Statistics - Week 16 (FU)
Description: Mean BSA score and change to baseline in treatment groups (150 and 300mg) compared to placebo at follow up visit. The BSA (Body Surface Area) provides information on the total surface area of the body affected with psoriasis plaques in percent (%).
Time Frame: Scoring took place on Site visits: Day1 (Baseline), Week 4, Week 8, Week 12 (End-of-Treatment), Week 16 (Follow-Up)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BSA (%)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 38 | 40 | 44
BSA (%)
  Week 16 (FU) | 20.9 (15.5) | 20.2 (19.8) | 15.5 (6.4)
  Week 16 (FU) - change from baseline | 0.6 (12.8) | 0.4 (13.4) | -1.1 (4.1)

38. Secondary Outcome: PK Data - Cmax
Description: The non-compartment parameter Cmax is the maximum MP1032 concentration observed based on the evaluation of systemic MP1032 concentrations in plasma samples wherein the respective blood samples were taken predose and 15, 30, 60 and 120 minutes after dosing.
Time Frame: Morning dose on Study Day 1
Population: The pharmacokinetics evaluation set (PKS) includes all patients without any protocol deviations that could have interfered with the administration of the treatment or the evaluation of systemic concentrations of MP1032, who received at least one dose of IMP and who had any completed determination of MP1032 levels.
Measure: Mean (Standard Deviation); unit: Cmax (ng/mL)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid
Number analyzed (Participants) | 6 | 8
Cmax (ng/mL) | 388 (146.3) | 612.4 (467.3)

39. Secondary Outcome: PK Data - Tmax
Description: The non-compartment parameter tmax is the time point (effective) at which the maximum concentration (Cmax) was observed based on the evaluation of systemic MP1032 concentrations in plasma samples wherein the respective blood samples were taken predose and 15, 30, 60 and 120 minutes after dosing.
Time Frame: Morning dose on Study Day 1
Population: as for outcome 38
Measure: Median (Full Range); unit: min
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid
Number analyzed (Participants) | 6 | 8
min | 15 [13 to 30] | 22.5 [15 to 60]

40. Secondary Outcome: PK Data - AUC(0,t)
Description: The non-compartment parameter AUC(0,t) is the area under the concentration-time curve up to the last quantifiable sample drawn based on the evaluation of systemic MP1032 concentrations in plasma samples wherein the respective blood samples were taken predose and 15, 30, 60 and 120 minutes after dosing.
Time Frame: Morning dose on Study Day 1
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: AUC(0,t) (ng/mL*min)
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid
Number analyzed (Participants) | 6 | 8
AUC(0,t) (ng/mL*min) | 15585.3 (5757.4) | 26543.8 (16592.3)

41. Secondary Outcome: Number of Patients With TEAEs
Description: Number of patients with treatment emergent adverse events (TEAEs) in treatment groups compared to placebo
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants | 22 | 15 | 33
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.1193, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0054, Fisher Exact

42. Secondary Outcome: Number of Patients With Serious TEAEs
Description: Number of patients with serious treatment emergent adverse events (TEAEs) in treatment groups compared to placebo
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants | 0 | 0 | 3
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.2439, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.2461, Fisher Exact

43. Secondary Outcome: Number of Patients With TEAEs Leading to Study Discontinuation
Description: Number of patients with treatment emergent adverse events (TEAEs) leading to study discontinuation in treatment groups compared to placebo
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants | 2 | 0 | 5
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.4395, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0593, Fisher Exact

44. Secondary Outcome: Number of Patients With TEAEs by SOC
Description: Number of patients with treatment emergent adverse events (TEAEs) in treatment groups compared to placebo displayed by MedDRA System Organ Classes (SOCs). Only PTs (MedDRA Preferred Terms) occuring in at least 5% of the patients were considered for this overview.
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants
  Infections and infestations | 11 | 8 | 14
  Skin and subcutaneous tissue disorders | 3 | 4 | 10
  Gastrointestinal disorder | 5 | 2 | 7
  Nervous system disorder | 2 | 4 | 2

45. Secondary Outcome: Number of Patients With TEAEs by Intensity
Description: Number of patients with treatment emergent adverse events (TEAEs) in treatment groups compared to placebo displayed by severity
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants
  Severe | 2 | 0 | 4
  Moderate | 7 | 4 | 15
  Mild | 13 | 11 | 14
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0507, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0005, Fisher Exact

46. Secondary Outcome: Number of Patients With TEAEs by Relation to the IMP
Description: Number of patients with treatment emergent adverse events (TEAEs) in treatment groups compared to placebo displayed according to investigators causality assessment.
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants
  Certainly related | 0 | 0 | 0
  Probably related | 1 | 0 | 1
  Possibly related | 4 | 2 | 8
  Unlikely related | 6 | 5 | 14
  Not related | 11 | 8 | 10
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0504, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0013, Fisher Exact

47. Secondary Outcome: Number of Patients With TEAEs by Causality With the IMP
Description: Number of patients with treatment emergent adverse events (TEAEs) in treatment groups compared to placebo displayed according to investigators causality assessment wherein "certainly", "probably" and "possibly related" were summarized as "related" whereas "unlikely" and "not related" were summarized as "not related".
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), Week 16 (Follow Up)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Number; unit: participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
participants
  Related | 5 | 2 | 9
  Not related | 17 | 13 | 24
Statistical Analysis 1: Comparison: 150 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.098, Fisher Exact
Statistical Analysis 2: Comparison: 300 mg MP1032 Bid vs Placebo Bid; Test type: Superiority; p = 0.0032, Fisher Exact

48. Secondary Outcome: Extent of Exposure - Dosed Capsules
Description: Total (cumulative) number of dosed capsules = 6 * # planned applications - # missed capsules + # overdose capsules.
  Planned were 2 applications (a 6 capsules) twice a day over a treatment period of 12 weeks. The number of missed and/or overdosed capsules is determined based on the restitution of used study drug packages.
Time Frame: overall trial / treatment period - cumulative from baseline to week 12 (EoT) or - if applicable - week16 (FU)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Mean (Standard Deviation); unit: capsules
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 47 | 55
capsules | 821.9 (304.3) | 920.6 (214.2) | 872.2 (248.3)

49. Secondary Outcome: Extent of Exposure - Capsules Per Application
Description: Average number of capsules per application = # dosed capsules / # applications.
  Planned were 2 applications (a 6 capsules) twice a day over a treatment period of 12 weeks. The number of missed and/or overdosed capsules is determined based on the restitution of used study drug packages.
Time Frame: overall trial / treatment period - from baseline to week 12 (EoT) or - if applicable - week16 (FU)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Mean (Standard Deviation); unit: capsules per application
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 47 | 55
capsules per application | 6.00 (0.02) | 6.00 (0.01) | 6.00 (0)

50. Secondary Outcome: Extent of Exposure - Capsules Per Day
Description: Average number of capsules per day = # dosed capsules / days of treatment.
  Planned were 2 applications (a 6 capsules) twice a day over a treatment period of 12 weeks. The number of missed and/or overdosed capsules is determined based on the restitution of used study drug packages.
Time Frame: overall trial / treatment period - from baseline to week 12 (EoT) or - if applicable - week16 (FU)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Mean (Standard Deviation); unit: capsules per day
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 47 | 55
capsules per day | 11.48 (1.40) | 11.85 (0.20) | 11.79 (0.20)

51. Secondary Outcome: Sufficient Extent of Exposure
Description: Exposure was regarded as sufficient if the patient took at least 80% of planned applications (respectively capsules) wherein % exposure was calculated as 100 * # dosed capsules / # planned capsules.
  Planned were 2 applications (a 6 capsules) twice a day over a treatment period of 12 weeks (i.e. 1008 capsules). The number of missed and/or overdosed capsules is determined based on the restitution of used study drug packages.
Time Frame: overall trial / treatment period - cumulative from baseline to week 12 (EoT) or - if applicable - week16 (FU)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 47 | 55
Participants
  Sufficient | 35 | 39 | 40
  Insufficient | 16 | 8 | 15

52. Secondary Outcome: Extent of Exposure - Treatment Duration
Description: Treatment duration = date of last dose - date of first dose + 1. 84 treatment days (12 weeks) were planned.
Time Frame: overall trial / treatment period - cumulative from baseline to week 4, 8, 12 (EoT), and - if applicable - week16 (FU)
Population: The safety-evaluation-set (SES) included all patients who received any trial medication at least once.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid
Number analyzed (Participants) | 51 | 48 | 55
days | 70.7 (24.1) | 76.1 (21.1) | 73.9 (21.0)

ADVERSE EVENTS:
Time Frame: Overall Trial - Explicit inquiry on Day1, Week 4, Week 8, Week 12 (EoT), and Week 16 (Follow Up). Additionally participants were encouraged to report AEs anytime between the visits.
Description: Only treatment-emergent AEs (TEAEs), i.e. AEs occuring after at least one dose of trial medication was administered, are listed in the investigational groups. All non treatment emergent AEs are listed in the screening/pretreatment column. AEs in the listing are described using the MedDRA Preferred Term (PT).
Groups:
- Screening / Pre-Treatment: This section includes all (non-treatment emergent) AEs that occured either in the screening phase (up to 28 days, overall 204 patients from whom eventually 155 patients were randomized to any of the intervention groups) or after randomization but before any IMP was administrated.
Arm/Group | 150 mg MP1032 Bid | 300 mg MP1032 Bid | Placebo Bid | Screening / Pre-Treatment
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48 | 0/55 | 0/204
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48 | 3/55 | 1/204
Other Adverse Events (participants affected / at risk) | 22/51 | 15/48 | 32/55 | 7/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg MP1032 Bid (N=51) | 300 mg MP1032 Bid (N=48) | Placebo Bid (N=55) | Screening / Pre-Treatment (N=204)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malum perforans (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg MP1032 Bid (N=51) | 300 mg MP1032 Bid (N=48) | Placebo Bid (N=55) | Screening / Pre-Treatment (N=204)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascariasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 5 (7) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Psoriasis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6) | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT03706209/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT03706209/SAP_001.pdf